CLINICAL TRIAL: NCT03565588
Title: Improving Risk Perception and Uptake of Voluntary Medical Male Circumcision (VMMC) With Education Sessions and Conditional Behavioural Incentives
Brief Title: Manicaland VMMC Uptake Through Behavioural Incentives Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Gregson (Other)
Collaborators: Biomedical Research and Training Institute, Zimbabwe (Other); University of Copenhagen (Other); London School of Economics and Political Science (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Simon Gregson, Professor of Demography and Behavioural Science, Imperial College London
Organization: Imperial College London (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P67251_VMMC; 1R01MH114562-01 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: HIV/AIDS
Keywords: Voluntary medical male circumcision; HIV prevention; Risk perception
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education session with fixed incentive (Experimental): Education sessions offered by a circumcised health worker and contribution towards transport costs to the health facility with payments conditional on being circumcised.
  Interventions: Behavioral: Education session with fixed incentive
- Education session with lottery incentive (Experimental): Education sessions offered by a circumcised health worker and contribution towards transport costs but with conditional lottery financial incentives.
  Interventions: Behavioral: Education session with lottery incentive
- Control arm (No Intervention): No intervention will be administered to the control arm

INTERVENTIONS:
Behavioral: Education session with fixed incentive — All participants will receive an education session on the risk of HIV infection and benefits from medical male circumcision. The sessions will be implemented by trained male healthcare workers who have undergone VMMC.
  All participants will receive contributions towards transport costs to access medical male circumcision at participating clinics. On completing VMMC, participants assigned to receive fixed incentives will receive payment through mobile payments. In two sites a community-led intervention will also be implemented to address social obstacles and to increase support from peers, families and social structures.
  Arms: Education session with fixed incentive
Behavioral: Education session with lottery incentive — All participants will receive an education session on the risk of HIV infection and benefits from medical male circumcision. The sessions will be implemented by trained male healthcare workers who have undergone VMMC.
  All participants will receive contributions towards transport costs to access medical male circumcision at participating clinics. On completing VMMC, participants will participate in a lottery with prizes equivalent in expected value to the fixed incentives. In two sites a community-led intervention will also be implemented to address social obstacles and to increase support from peers, families and social structures.
  Arms: Education session with lottery incentive

SUMMARY:
Primary Objective The purpose of this study is to evaluate the impact of an interactive VMMC education session offered by a circumcised health worker and contribution to transport costs for accessing VMMC along with either (1) conditional economic compensation for wages or (2) lottery-based economic incentives on the uptake of VMMC.

Hypothesis VMMC education session offered by a role model - a young male health worker who has been previously benefited from VMMC services in this community - addressing risks of HIV infection, benefits of VMMC, and the fear of pain associated with VMMC, with/without a conditional fixed or lottery-based financial incentives off-setting present-biased preferences, will improve risk perception and increase uptake of VMMC in HIV-negative young men.

Study outcomes The primary outcomes for the study will be risk perception measured in a follow-up survey at 6 months and proportion of men taking up VMMC within 6 months measured through self-reports and matched to program records.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 15-29 years

Exclusion Criteria:

* Participants testing HIV-positive at baseline
* Self-reporting have already undergone circumcision

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 1028 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Uptake of voluntary medical male circumcision (VMMC) | 6 months
  Proportion of men taking up VMMC within 6 months measured through self-reports and matched to programme records

SECONDARY OUTCOMES:
Changes in perception of risk of HIV | 6 months
  Risk perception will be measured in a follow-up survey at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gregson, PhD, Principal Investigator — Imperial College London
Locations (7):
- Zimbabwe (7):
  - Manicaland Centre for Public Health Research, Bonda, Manicaland Province
  - Manicaland Centre for Public Health Research, Hobhouse, Manicaland Province
  - Manicaland Centre for Public Health Research, Honde, Manicaland Province
  - Manicaland Centre for Public Health Research, Manicaland, Manicaland Province
  - Manicaland Centre for Public Health Research, Nyanga, Manicaland Province
  - Manicaland Centre for Public Health Research, Nyazura, Manicaland Province
  - Manicaland Centre for Public Health Research, Sakubva, Manicaland Province

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thomas R, Skovdal M, Galizzi MM, Schaefer R, Moorhouse L, Nyamukapa C, Maswera R, Mandizvidza P, Hallett TB, Gregson S. Improving risk perception and uptake of voluntary medical male circumcision with peer-education sessions and incentives, in Manicaland, East Zimbabwe: study protocol for a pilot randomised trial. Trials. 2020 Jan 23;21(1):108. doi: 10.1186/s13063-020-4048-2. PMID 31973744